CLINICAL TRIAL: NCT01319019
Title: A 4-week Dose-Ranging, Dose-Interval, Efficacy, Safety and Tolerability Study of GSK961081 in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115032
Record Dates: First submitted 2011-03-03; First posted 2011-03-21 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: lung function; bronchodilator; COPD, dose response, dosing interval, efficacy, safety, PD, PK
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — batefenterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- GSK961081 100 mcg QD (Experimental)
  Interventions: Drug: GSK961081
- GSK961081 100mcg BD (Experimental)
  Interventions: Drug: GSK961081
- GSK961081 200mcg QD (Experimental)
  Interventions: Drug: GSK961081
- GSK961081 400mcg QD (Experimental)
  Interventions: Drug: GSK961081
- GSK961081 400mcg BD (Experimental)
  Interventions: Drug: GSK961081
- GSK961081 800mcg QD (Experimental)
  Interventions: Drug: GSK961081
- Salmeterol 50mcg BD (Active Comparator)
  Interventions: Drug: Salmeterol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK961081 — Comparison of different doses and dosing regimens of the drug
  Arms: GSK961081 100 mcg QD; GSK961081 100mcg BD; GSK961081 200mcg QD; GSK961081 400mcg BD; GSK961081 400mcg QD; GSK961081 800mcg QD
Drug: Salmeterol — Positive control
  Arms: Salmeterol 50mcg BD
Drug: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
This study is primarily designed to assess the dose response, dose interval, efficacy and safety of three once daily (QD) doses (100mcg, 400mcg and 800mcg) and three twice daily (BID) doses (100mcg, 200mcg and 400mcg,) of GSK961081 administered via DISKUS™ for 28 days in subjects with moderate/severe COPD versus placebo. Salmeterol 50mcg BID is included in the study as an active comparator.

DETAILED DESCRIPTION:
This is a phase IIb multicentre, randomised, double-blind, double-dummy, placebo- and active-controlled, parallel-group, dose-ranging and dose-interval study. Eligible subjects will enter a seven-day run-in period followed by 28 days of double-blind, double-dummy treatment via the DISKUS inhaler. The study will consist of 8 visits, mainly conducted on an outpatient basis, 6 of which will be clinic visits and 2 of which will be phone contacts, including a post-treatment visit to follow up any adverse events. There will be approximately 425 subjects randomised to the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient Subjects
* Subjects who give their signed and dated informed consent to participate
* 40 or more years of age, inclusive, at Visit 1
* Male or females
* Subjects with an established clinical history of COPD
* Current or previous cigarette smokers with a history of ≥ 10 pack-years of cigarette smoking
* Subjects with the following liver function test values:
* Subjects with a measured post-salbutamol FEV1/FVC ratio of < 0.70 at Visit 1 (Screening).
* Subjects with a measured post-salbutamol FEV1 30-70% of predicted normal values

Exclusion Criteria:

* Women who are pregnant or lactating or are planning to become pregnant during the study.
* Current diagnosis of asthma
* Other significant respiratory disorders besides COPD, including alpha-1 deficiency
* Previous lung resection surgery
* Significant abnormalities in chest x-ray presentation
* Hospitalization for a COPD exacerbation within 12 weeks prior screening
* Use of oral corticosteroids or antibiotics for COPD or antibiotics for a lower respiratory tract infection within 6 weeks
* Any significant disease that would put subject at risk through study participation
* BMI greater than 35
* Pacemaker
* Significantly abnormal ECG, clinical lab finding (including Hepatitis B or C)
* Cancer
* Allergy or hypersensitivity to beta adrenergic receptor-agonist, sympathomimetic, anticholinergic/anti-muscarinic receptor antagonist, or inhaler excipients
* Diseases that would contra-indicate the use of anticholinergics
* Use of sysemic corticosteroids within 6 weeks of screening
* Use of long-acting beta-agonists within 48 hours of screening
* Use of tiotropium within 7 days of screening
* Use of theophyllines or anti-leukotrienes within 48 hours of screening
* Use of short-acting bronchodilators within 4 hours of screening
* Use of investigational medicines within 30 days of screening
* Use of high dose inhaled corticosteroids
* Use of long-term oxygen therapy, CPAP or NIPPV
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1
* Regular (q.i.d or greater) use of short acting bronchodilators, including nebulized therapy
* Affiliation with Investigator Site
* Questionable Validity of Consent
* Previous use of GSK961081

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 from baseline in pre-dose AM trough. | 28 Day
  Pre-dose change in AM FEV1 on day 29 vs baseline . (defined as the mean values recorded 11 and 12 hours after the PM dose on day 28)

SECONDARY OUTCOMES:
Weighted Mean and Serial FEV1 at multiple timepoints | 28 Days
  In the subset of patients with overnight spirometry on day 28 (pre-dose and post dose after 15,30, and 60 min and 2, 4,6, 11 and 12 hours)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (5):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Netherlands (6):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zutphen
- Romania (3):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Timișoara
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yekaterinburg
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Zámky
  - GSK Investigational Site, Zvolen
- South Africa (6):
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Gatesville
  - GSK Investigational Site, Mowbray
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Tygerberg
- Sweden (4):
  - GSK Investigational Site, Boden
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Wielders PL, Ludwig-Sengpiel A, Locantore N, Baggen S, Chan R, Riley JH. A new class of bronchodilator improves lung function in COPD: a trial with GSK961081. Eur Respir J. 2013 Oct;42(4):972-81. doi: 10.1183/09031936.00165712. Epub 2013 Feb 21. PMID 23429913
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115032 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register